CLINICAL TRIAL: NCT03231163
Title: Physiological and Perceptual Effects of Music on Resting Metabolic Rate (RMR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Assistant Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1082672-3
Record Dates: First submitted 2017-07-23; First posted 2017-07-27 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Music (Placebo Comparator)
  Interventions: Other: No Music
- Relaxing Classical Music (Experimental)
  Interventions: Other: Relaxing Classical Music
- Self-Selected Relaxing Music (Experimental)
  Interventions: Other: Self-Selected Relaxing Music

INTERVENTIONS:
Other: No Music — Participants lie supine on a table while no music is played.
  Arms: No Music
Other: Relaxing Classical Music — Participants lie supine on a table while classical music is played.
  Arms: Relaxing Classical Music
Other: Self-Selected Relaxing Music — Participants lie supine on a table while self-selected relaxing music is played.
  Arms: Self-Selected Relaxing Music

SUMMARY:
The objective of the study is to determine whether music has any effect on resting metabolic rate (RMR), which is the amount of energy expended at rest. There is currently conflicting research on how music affects RMR. One problem with RMR testing is that participants often fall asleep during the test. There can be a 5-10% difference in the metabolic rate between rest and sleep. If no change in RMR is observed, playing music during an RMR test could be a potential strategy to prevent participants from falling asleep. Participants will undergo RMR measurements while listening to no music, relaxing classical music, and self-selected classical music.

ELIGIBILITY:
Exclusion Criteria:

* Any metabolic disorder, or significant cardiopulmonary disease
* Taking medications that are known to affect RMR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Daily Resting Metabolic Rate | Participants will be randomized to three consecutive 15-minute trials involving listening to no music, classical music, or self-selected relaxing music. RMR will be measured continuously over each 15 min trial.
  RMR will be measured via indirect calorimetry (Parvomedics TrueOne system)

SECONDARY OUTCOMES:
Heart rate | Participants will be randomized to three consecutive 15-minute trials involving listening to no music, classical music, or self-selected relaxing music. Heart rate will be measured continuously over each 15 min trial.
  Heart rate will be measured with a Polar chest strap monitor
Excited/bored scale | Participants will be randomized to three consecutive 15-minute trials involving listening to no music, classical music, or self-selected relaxing music. Levels of boredom/excitement will be measured at the end of each 15 min trial.
  Participants rate on a 0-9 Likert scale how bored or excited they are.
Sleepiness scale | Participants will be randomized to three consecutive 15-minute trials involving listening to no music, classical music, or self-selected relaxing music. Levels of sleepiness will be measured at the end of each 15 min trial.
  Participants rate on a 0-9 Likert scale how sleepy they are.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No